CLINICAL TRIAL: NCT00561704
Title: Adiponectin in Obese Women With T2DN and Effects by RAS Blocker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADL
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Obese; Type 2 Diabetes; Diabetic Nephropathy; Glucose Metabolism; Angiotensin II Type 1 Receptor Blockers
Keywords: obese female; Type 2 Diabetes; Diabetic Nephropathy; Glucose Metabolism; Angiotensin II Type 1 Receptor Blockers; Adiponectin
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: losartan — losartan, 100mg daily,

SUMMARY:
Insulin resistance typically characterizes type 2 diabetes (T2DM) and prediabetic states and is the prominent feature of the metabolic syndrome.Adiponectin plays an important part in glucose metabolism,insulin resistance, the deterioration of renal function.we hypothesize there is a difference serum adiponectin levels between obese and non-obese women with type 2 diabetic nephropathy. Furthermore, these two groups would respond difference to the RAs blocker(Losartan).

DETAILED DESCRIPTION:
it would be a prospective cohort study. According to BMI, all the women, aged>30yr, diagnosed type 2 diabetic nephropathy, chronic kidney disease stage range from 1 to 4, will be divided to two group. Renal function index(included SCr, GFR, et al),glucose metabolism index( fasting glucose, plasma insulin et al),and adiponectin concentration will be observed and recorded. both two groups females will accept the treatment of RAS blocker(losartan, 100mg daily, 6 month). during the study, the above mentioned parameters will also be recorded 3 month intervals. Meanwhile, any side effects would be pay attention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic nephropathy
* CKD at stage 1~4

Exclusion Criteria:

* Type 1 diabetes or nondiabetic renal disease
* An elevated plasma K level.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
GFR, HbA1c and the adiponectin concentration. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: hui min Jin, MD, Principal Investigator — shanghai No 3 people's hospital